CLINICAL TRIAL: NCT07139808
Title: Safety and Effectiveness of A Novel Continuous Glucose and Ketone Monitoring System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Peng Liu, Investigator, Henan University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SS-KY-CGM-0004
Record Dates: First submitted 2025-08-15; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with T1DM (Experimental): Adult patients with T1DM
  Interventions: Device: GK5 CGKM

INTERVENTIONS:
Device: GK5 CGKM — Wear for a consecutive 15 days

SUMMARY:
The study is to evaluate the accuracy and safety of a novel real-time continuous glucose and ketone monitoring system among adult patients with type 1 diabetes mellitus (T1DM) with respect to Yellow Spring Instrument (YSI) and Randox reference venous plasma sample measurements.

DETAILED DESCRIPTION:
The study is to evaluate the accuracy and safety of a novel real-time continuous glucose and ketone monitoring (CGKM) system among adult patients with type 1 diabetes mellitus with respect to YSI and Randox reference venous plasma sample measurements. Up to 14 patients will be enrolled. Interstitial glucose and ketone readings from the sensors will be obtained immediatedly following each venous blood sample test. Each participant will make 3 visits to the clinical study site, including the screening visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagonsed with T1DM on Continuous subcutaneous insulin infusion (CSII)
* Venous blood sampling access can be established in the forearm
* Capable of independently reading instructions and complying with the clinical trial requirements
* Willing to sign the Informed Consent Form (ICF)

Exclusion Criteria:

* Severe hypoglycemia within the past 6 months
* A diagnosed history of Diabetic ketoacidosis (DKA) in the past 3 months
* Heart failure or hemiplegic sequelae due to prior cerebrovascular disease
* Severe skin conditions at the sensor wear site
* Extensive systemic skin disorders
* Having difficulty with wound healing, bleeding disorders, and/or taking anticoagulant medications
* Anemia or abnormal hematocrit
* Blood donation within the past 6 months
* Pregnancy (defined as positive urine test in women ≤55 years), lactation, or plans for pregnancy within ≤30 days
* Current or recent (≤1 month) participation in other clinical trials
* Planned MRI/CT scans during sensor wear
* Allergy to medical adhesives or alcohol
* Conditions impairing comprehension of informed consent or study procedures
* Other exclusionary conditions per investigator's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
System performance on glucose measurement | 15 days
  The CGK system performance for glucose measurement will be assessed by comparing to the Yellow Springs Instrument comparator venous plasma measurements
System performance on ketone measurement | 15 days
  The CGK system performance for ketone measurement will be assessed by comparing to the Randox comparator venous plasma measurements

SECONDARY OUTCOMES:
System-related Safety | 15 days
  Records of the adverse events and device-related incidence rates.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Jiang, Principal Investigator — Henan University of Science and Technology
Locations (1):
- Henan University of Science and Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No